CLINICAL TRIAL: NCT02938676
Title: Satisfaction Degree With the Education Received in an Educational Program to Heart Transplant Patient During Hospitalization
Brief Title: Satisfaction Degree in a Nurse Educational Program to Heart Transplant Patient
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Other Study IDs: IIBSP-SAT-2016-44
Record Dates: First submitted 2016-10-10; First posted 2016-10-19 (Estimated); Last update posted 2016-10-19 (Estimated); Status verified 2016-10

CONDITIONS: Heart Transplantation; Health Education
MeSH Terms: conditions — Health Education

STUDY DESIGN:
Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Any member of the research team conducted screening for the selection of eligible patients. Nurses will be responsible for delivering the "Guide tips for the person with a transplanted heart", thus initiating an individualized education program. Education will be held at the time of admission in which the patient has passed the most critical post-operative.

Educational tips guide contains all the information necessary for the patient to have a first contact on the habits that must change. Education lasts 10-30 minutes and is taught in daytime, in a calm environment and at the right time, favoring the presence of the caregiver. Later, education is reinforced on the doubts that arise both the patient and the primary caregiver.

During the first days of admission to the unit of cardiology, socio-demographic data of the patient and primary caregiver by the research team will be collected.

A few days before discharge, having left time between 7-8 days after delivery of educational advice guide, any member of the research team, who does not work in the cardiology unit, will provide the patient and the primary caregiver the satisfaction questionnaire where the perception of information and education received during the postoperative period in the inpatient cardiology unit and the appropriateness of the topics covered in the guide educational advice.

DETAILED DESCRIPTION:
* Conceptual Definition: Result of the difference between what the patient / caregiver expected to happen (patient expectations) and what claims to have obtained (their perception of the experience, the service provided) 14, 15.
* Operational Definition: To assess the degree of satisfaction has designed a self-administered questionnaire specific for this study in which the following items were evaluated:

  1. Knowledge of the name and profession of the person performing the educational activity.
  2. Time used to provide educational session.
  3. Adequacy of time spent by nurses.
  4. At which has been given the educational session.
  5. Educational information received.
  6. Documentation provided.
  7. Understanding the information provided.
  8. Specific content by topics (general information, diet, hygiene measures, mood, exercise and cardiac rehabilitation, sexual activity, complications, skin, eye, gastrointestinal tract, bones, toxic habits, vaccination, contact other people, animals and plants, travel, employment high, associations heart transplant recipients).
  9. Satisfaction with education received

The overall satisfaction score is obtained from the sum of the scores of all items and a cut will be established from data obtained from median scores in a previous pilot survey conducted using 5 patients. The overall satisfaction score can range from 0 to 120 points.

ELIGIBILITY:
Inclusion Criteria:

* Patients of both sexes, over 18 years.
* With medical diagnosis of heart transplant surgery during the same hospitalization.
* They must have a "primary caregiver" or a report favorable social support.

Exclusion Criteria:

* Medical diagnosis of cognitive impairment (Alzheimer's disease, senile dementia, neurological problem).
* Illiteracy and / or language barrier.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients Unit hospitalization of Cardiology (B3) of the Hospital de la Santa Creu i Sant Pau (HSCSP) that during admission require surgery Heart Transplantation.
  Convenience sampling in which eligible patients will be selected to participate in the study consecutively according to the time of admission to the inpatient
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2016-11; Primary Completion 2018-01 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Patient satisfaction by a a self-administered questionnaire specific to this study | 1 year
  It will be evaluated:
  1. Knowledge of the name and profession of the person performing the educational activity.
  2. Time used to provide educational session.
  3. Adequacy of time spent by nurses.
  4. At which has been given the educational session.
  5. Educational information received.
  6. Documentation provided.
  7. Understanding the information provided.
  8. Specific content by topics
  9. Satisfaction with education received in general The overall satisfaction score is obtained from the sum of the scores of all items and a cut will be established from data obtained from median scores in a previous pilot survey conducted using 5 patients. The overall satisfaction score can range from 0 to 120 points.

CONTACTS AND LOCATIONS:
Overall Officials: Alba Villalobos Abelló, Principal Investigator — Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau

IPD SHARING:
Plan to Share IPD: Undecided